## Effects of Blood Orange Juice Consumption on Endothelial Function in Healthy Overweight/Obese Men and Premenopausal Women of European Origin

Date: January 10, 2017

Statistical analysis will be conducted by using Statistical Package for the Social Sciences (SPSS, version 24, IBM Corporation, USA). Data will be tested for normality by using Shapiro-Wilk test. Data at the end of each treatment will be analysed by using a linear mixed model for crossover trials, with age, BMI, baseline values as covariates, subjects nested within treatment sequence as the random effect, and gender, dietary treatment, treatment sequence, experimental period, the interaction between treatment and experimental period as fixed effects. Significance is defined at p < 0.05. Pearson's correlation analyses will be conducted.